## **Official Title:** Reengaging rural patients in VA mental health care after VA-community care network referral

NCT Number: NCT06139887

**Document Date:** 01/02/2024

## **Telephone Consent Script for BESST RCT**

**Study Title:** Reengaging rural patients in VA mental health care after VA-community care network referral

**IRB#:** 1701666

Name of person conducting the consent:

## **Introduction:**

Hello, is this [insert name of Veteran]? My name is [insert name of study staff member] from the White River Junction VA Medical Center. I am following up on a letter and information sheet my team and I sent you describing our research study on a program called the <u>Building VA Engagement</u>, <u>Self-Efficacy</u>, and <u>Social Support To Prevent Suicide or the "BESST" program. My team and I are studying the BESST program to see if it helps Veterans maintain involvement in mental health care and enhance their sense of social connectedness with others. Dr. Natalie Riblet of the White River Junction VA runs this study. If you are interested in hearing more, I'd like to tell you more about the study and see if you might want to participate.</u>

Would you like to hear more about the study?

Yes

No

We are asking you to be in this study because you are a patient of [insert VA medical center] and have received care at a community care site. For you, that was [insert type of setting, e.g., mental health hospitalization]. The purpose of this study is to learn if the BESST program can help Veterans who are discharged from community care sites. Veterans with mental health symptoms may be at higher risk for suicidal thoughts and behaviors. This risk can be caused by many things, including challenges in accessing mental health care and low feelings of social connectedness. So, we are studying the BESST program to see if it can help Veterans remain involved with their care and prevent suicide. We specifically want to study the BESST program among Veterans who have received community care because more and more Veterans are receiving treatment in these settings.

Your participation in this study is voluntary with minimal risk to you. Your decision about being in this study will have no effect on you or your health care in the VA. If you decline to enter the study, there will be no penalty or loss of benefits to which you are otherwise entitled to. You can choose to withdraw from this study at any time. Please feel free to ask questions if there is any information you do not understand.

Version: 1.2.2024

Before I ask your consent to participate, I'd like to explain what information we will collect and how we will store it. We will make every effort to protect your identity and the confidentiality of the data collected. For example, the information we collect remains on a secure VA folder, which only certain research staff can access using their unique login information. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

If you decide to join this study, you will be assigned by chance to a treatment group. Some will be in the group that receives the BESST program, and some will be in the group that receives standard mental health treatment. Standard mental health treatment simply refers to the regular care provided to you around the time of discharge from community care. If assigned to receive the BESST program, you would be in this research for up to three months and participate in eight study visits as well as three study interviews. All BESST program visits can be completed over phone, VVC, or in-person based on your preference. If you would prefer to have your study visits in-person, you will need to ensure reliable transportation to the White River Junction VA Medical Center campus. The BESST program includes a one-hour brief educational session and seven follow-up check-ins that will take approximately 30 minutes. The brief educational session will include information on suicide prevention, a discussion of your mental health care after discharge, and a review of helpful resources. During the check-ins, our study provider will work with you to help you stay connected to your regular treatment providers.

If you are assigned to the group that receives standard mental health care, you would also be in this study for up to three months and participate in three study interviews.

The three study interviews will be completed by all participants from both groups. During these visits, we will ask you a set of standardized questions about your mental health and if you received any treatment outside of the VA during the study. The first study interview will occur around the time of discharge and takes approximately 1 hour. Follow-up study interviews occur at one- and three-months after the first interview and take approximately 30 minutes. These visits can be completed over the phone or VVC. At the end of the three months, study staff will look in your medical chart to record any treatment you received within the VA during the study.

For all visits completed over the phone or VVC, we ask that you are in a location where you feel safe and comfortable. For your safety, we also ask that you do not drive a vehicle while participating in study visits.

Finally, if you enroll in the study, you will be paid up to \$300 for your time and effort. The payment will be provided to you as a direct deposit into your bank account. You will receive \$100 for each completed assessment, for a total of \$300. You can decide to either receive a lump sum at the end of your time in the study or receive payment after completion of each assessment. If you decide to discontinue before completing all study visits, you will be compensated for the assessments that you did complete.

Version: 1.2.2024

| Do you have any questions about the study? (if none, write "none" below). |
|---|
| Your verbal consent means that you understand the information I shared with you and that you agree to take part in this study. Do you agree to participate in this research study? Yes No |
| Thank you for agreeing to participate in this study. I would like to give you some phone numbers in case you have some questions about this study in the future. Please call Dr. Natalie Riblet at 802-299-8682 during normal business hours if you have a specific question about the study. If you have questions, concerns, complaints, or suggestions about human subjects research at the White River Junction VA Medical Center, you can call the office for the Veteran's Institutional Review Board of Northern New England (VINNE) at 802-295-9363 x5837 during normal business hours. |
| *Complete after verbal consent is obtained: |
| Name of Veteran: |
| Last 4 SSN: |
| Date of Consent: |
| Time of Consent: |

Version: 1.2.2024